CLINICAL TRIAL: NCT00660036
Title: Phase I/II Study of the Combination of Mitoxantrone, Etoposide and Gemtuzumab Ozogamicin for Patients With Acute Myeloid Leukemia Refractory to Initial Standard Induction Therapy (UPCI 07-154)
Brief Title: Phase I/II Study of Mitoxantrone, Etoposide and Gemtuzumab Ozogamicin for Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: due to new safety information
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Michael Boyiadzis, PI, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-154
Record Dates: First submitted 2008-04-11; First posted 2008-04-17 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Refractory; Relapsed; Second line; Gemtuzumab ozogamicin; Mitoxantrone; Etoposide; Phase I; Phase II
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Gemtuzumab; Mitoxantrone; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemtuzumab ozogamicin/Mitoxantrone/Etoposide (Experimental)
  Interventions: Drug: Gemtuzumab ozogamicin; Drug: Mitoxantrone; Drug: Etoposide

INTERVENTIONS:
Drug: Gemtuzumab ozogamicin — On Day 6 of an inpatient hospital stay: Based on the study design patients will be treated with one of three doses (3 mg/m^2, 6 mg/m^2 or 9 mg/m^2), administered intravenously in 100 ml of 0.9% sodium chloride over 2 hours.
  Other Names: Mylotarg®
Drug: Mitoxantrone — On Days 1-3 of an inpatient hospital stay: 10 mg/m^2 administered via IVPB (intravenous piggy-back) in 50ml normal saline (NS) over 15 minutes
  Other Names: Novantrone®
Drug: Etoposide — On Days 1-5 of an inpatient hospital stay: 100 mg/m^2 administered intravenously in 500 ml of 0.9% sodium chloride over 2 hours
  Other Names: ToposarTM

SUMMARY:
The purpose of this study is to investigate the combination of gemtuzumab ozogamicin, mitoxantrone and etoposide as second line therapy in patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
The combination of mitoxantrone and etoposide is an active regimen in refractory/relapsed AML patients. In order to improve the efficacy of mitoxantrone and etoposide as second line therapy in patients with AML we proposed to conduct a phase I/II clinical trial combining gemtuzumab ozogamicin with mitoxantrone and etoposide. The phase I portion of the trial will determine the maximum tolerated dose of gemtuzumab ozogamicin combined with mitoxantrone and etoposide and the phase II portion of the trial will determine the efficacy and safety of the combined regimen in patients with AML.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and have the ability to provide written consent
* Between 18 and 70 years of age
* Patients with CD33 positive (determined as CD33 expression in ≥ 20% of leukemic blasts) de novo AML that did not respond to first line induction therapy
* ECOG Performance Status of 0-2
* Patients must have the following laboratory values within 48 hours prior to beginning protocol treatment: Serum creatinine ≤ 1.5 mg/ml and calculated creatinine clearance ≥ 50mL/min (using the Cockcroft-Gault equation); AST ≤ 59 IU/L; ALT ≤ 72 IU/L; Total bilirubin ≤ 1.3 mg/ml; Note: Hematologic abnormalities will not be used as a criteria for entry or exclusion.
* Patients must have left ventricular ejection fraction (LVEF) ≥50%
* Females of child-bearing potential must have a negative pregnancy test during screening and all subjects must agree to use an effective method of contraception.

Exclusion Criteria:

* Patients with acute promyelocytic leukemia
* Prior use of mitoxantrone or etoposide or gemtuzumab ozogamicin
* Antecedent hematologic disorder preceding initial presentation of AML or therapy related AML
* History of thromboembolic event within the past 12 months
* Hepatitis B or C or HIV positive serology
* Symptomatic central nervous system (CNS) involvement
* History of congestive heart failure
* Myocardial infarction in the past 6 months
* Uncontrolled, life-threatening infection that is not responding to antimicrobial therapy
* History of psychiatric disorder which may compromise compliance with the protocol or which does not allow for appropriate informed consent
* Patient may not be receiving any other anti neoplastic investigational agents
* INR> 1.5 or patient is receiving systemic anticoagulation (e.g warfarin)
* Patient undergone autologous or allogeneic stem cell transplantation
* Other active malignancies except for non-melanoma skin cancer or cervical intraepithelial neoplasia
* Women who are pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the toxicity and response rate of the combination therapy of mitoxantrone, etoposide and gemtuzumab ozogamicin as second line therapy in patients with acute myeloid leukemia (AML). | Bone marrow biopsy and aspiration 14 days after gemtuzumab ozogamicin administration, to evaluate response to the study drug regimen.

SECONDARY OUTCOMES:
To assess the overall survival in patients with AML treated with the combination of mitoxantrone, etoposide and gemtuzumab ozogamicin. | Indefinite; subjects are followed for survival.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boyiadzis, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute / Hillman Cancer Center, Pittsburgh, Pennsylvania, United States